CLINICAL TRIAL: NCT06506812
Title: Pooled Analysis of Methodologically Harmonized Pragmatic Randomized Trials of High-Dose vs. Standard-Dose Influenza Vaccine Against Severe Clinical Outcomes
Acronym: FLUNITY-HD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tor Biering-Sørensen (Other)
Collaborators: Sanofi (Industry); Hospital Clinico Universitario de Santiago (Other)
Responsible Party: Sponsor-Investigator, Tor Biering-Sørensen, Professor, MD, MSc, MPH, PhD, Herlev and Gentofte Hospital
Organization: Herlev and Gentofte Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DANFLU/GALFLU pooled analysis
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Influenza
Keywords: Influenza; Vaccination; Pragmatic; Registry; Pneumonia; Respiratory; Cardiovascular; Meta-analysis
MeSH Terms: conditions — Influenza, Human; Pneumonia | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Dose Influenza Vaccine (Experimental): Single injection of high-dose influenza vaccine at Day 0
  Interventions: Biological: High-Dose Influenza Vaccine
- Standard-Dose Influenza Vaccine (Active Comparator): Single injection of standard-dose influenza vaccine at Day 0
  Interventions: Biological: Standard-Dose Influenza Vaccine

INTERVENTIONS:
Biological: High-Dose Influenza Vaccine — For this arm, the high-dose quadrivalent influenza vaccine Efluelda®/Fluzone® High-Dose Quadrivalent will be used.
  Arms: High-Dose Influenza Vaccine
Biological: Standard-Dose Influenza Vaccine — Any standard-dose quadrivalent influenza vaccine administered in the governmental influenza vaccine programs may be used.
  Arms: Standard-Dose Influenza Vaccine

SUMMARY:
This prespecified analysis will pool the datasets from two pragmatic randomized trials evaluating the relative vaccine effectiveness of high-dose vs. standard-dose influenza vaccine against severe clinical outcomes: the DANFLU-2 (A Pragmatic Randomized Trial to Evaluate the Effectiveness of High-Dose Quadrivalent Influenza Vaccine vs. Standard-Dose Quadrivalent Influenza Vaccine in Older Adults) trial and the GALFLU (Pragmatic Randomized Trial to Evaluate the Effectiveness of High-Dose Quadrivalent Influenza Vaccine vs. Standard-Dose Quadrivalent Influenza Vaccine in Adults Aged 65 to 79 Years in Galicia, Spain) trial. The purpose of the pooled analysis is to ensure adequate statistical power for evaluating relative vaccine effectiveness against severe clinical outcomes and to increase generalizability of the results by combining data from two countries.

ELIGIBILITY:
Inclusion Criteria:

* Pragmatic trials conducted to estimate the relative vaccine effectiveness of high-dose influenza vaccine compared with standard-dose influenza vaccine using the DANFLU-2 protocol or a protocol developed based on the DANFLU-2 protocol

Exclusion Criteria:

* Low data quality
* Influenza circulation threshold was not met in any of the study seasons
* Severe under-enrollment in all seasons

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 466320 (Actual)
Dates: Start 2025-05-31 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Hospitalization for influenza or pneumonia | ≥14 days after vaccination up to 8 months

SECONDARY OUTCOMES:
Hospitalization for any cardio-respiratory disease | ≥14 days after vaccination up to 8 months
Laboratory-confirmed influenza hospitalization | ≥14 days after vaccination up to 8 months
All-cause hospitalization | ≥14 days after vaccination up to 8 months
All-cause mortality | ≥14 days after vaccination up to 8 months
Hospitalization for influenza | ≥14 days after vaccination up to 8 months
Hospitalization for pneumonia | ≥14 days after vaccination up to 8 months

OTHER OUTCOMES:
Hospitalization for influenza or pneumonia (alternate definition) | ≥14 days after vaccination up to 8 months
Hospitalization for pneumonia (alternate definition) | ≥14 days after vaccination up to 8 months
Hospitalization for influenza (alternate definition) | ≥14 days after vaccination up to 8 months
Hospitalization for any respiratory disease | ≥14 days after vaccination up to 8 months
Hospitalization for any cardiovascular disease | ≥14 days after vaccination up to 8 months
Hospitalization for myocardial infarction | ≥14 days after vaccination up to 8 months
Hospitalization for heart failure | ≥14 days after vaccination up to 8 months
Hospitalization for atrial fibrillation | ≥14 days after vaccination up to 8 months
Hospitalization for stroke | ≥14 days after vaccination up to 8 months
Major adverse cardiovascular events (MACE) defined as a composite of hospitalization for acute myocardial infarction, hospitalization for stroke, and cardiovascular death | ≥14 days after vaccination up to 8 months
MACE defined as a composite of hospitalization for acute myocardial infarction, hospitalization for stroke, hospitalization for heart failure, and cardiovascular death (alternate definition #1) | ≥14 days after vaccination up to 8 months
MACE defined as a composite of hospitalization for acute myocardial infarction, hospitalization for stroke, and all-cause death (alternate definition #2) | ≥14 days after vaccination up to 8 months
Hospitalization requiring mechanical ventilation | ≥14 days after vaccination up to 8 months
Laboratory-confirmed influenza | ≥14 days after vaccination up to 8 months
Laboratory-confirmed pneumococcal pneumonia | ≥14 days after vaccination up to 8 months
Laboratory-confirmed COVID-19 | ≥14 days after vaccination up to 8 months
Cardio-respiratory mortality | ≥14 days after vaccination up to 8 months
Respiratory mortality | ≥14 days after vaccination up to 8 months
Cardiovascular mortality | ≥14 days after vaccination up to 8 months
In-hospital mortality | ≥14 days after vaccination up to 8 months
Intensive care unit admission | ≥14 days after vaccination up to 8 months
Any hospital contact associated with laboratory-confirmed influenza | ≥14 days after vaccination up to 8 months
Any exacerbation of pre-existing chronic obstructive pulmonary disease | ≥14 days after vaccination up to 8 months
Any exacerbation of pre-existing chronic obstructive pulmonary disease (alternate definition) | ≥14 days after vaccination up to 8 months
Severe exacerbation of pre-existing chronic obstructive pulmonary disease | ≥14 days after vaccination up to 8 months
Severe exacerbation of pre-existing chronic obstructive pulmonary disease (alternate definition) | ≥14 days after vaccination up to 8 months
Any exacerbation of pre-existing asthma | ≥14 days after vaccination up to 8 months
Any exacerbation of pre-existing asthma (alternate definition) | ≥14 days after vaccination up to 8 months
Severe exacerbation of pre-existing asthma | ≥14 days after vaccination up to 8 months
Severe exacerbation of pre-existing asthma (alternate definition) | ≥14 days after vaccination up to 8 months
Exacerbation of pre-existing heart failure | ≥14 days after vaccination up to 8 months
Exacerbation of pre-existing heart failure (alternate definition) | ≥14 days after vaccination up to 8 months
Hospitalization for pericarditis | ≥14 days after vaccination up to 8 months
Hospitalization for myocarditis | ≥14 days after vaccination up to 8 months
New-onset dementia | ≥14 days after vaccination up to 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Tor Biering-Sørensen, MD, MSc, MPH, PhD, Study Chair — Center for Translational Cardiology and Pragmatic Randomized Trials, Department of Cardiology, Copenhagen University Hospital - Herlev and Gentofte
Locations (1):
- Center for Translational Cardiology and Pragmatic Randomized Trials, Department of Cardiology, Copenhagen University Hospital - Herlev and Gentofte, Hellerup, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Yes
In each trial, baseline and endpoint data will be collected from administrative health registries, which are subject to local legislation and can only be made available to a third party under certain conditions. Please contact the sponsor in case of any inquiries.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Johansen ND, Modin D, Pardo-Seco J, Rodriguez-Tenreiro-Sanchez C, Loiacono MM, Harris RC, Dufournet M, van Aalst R, Chit A, Larsen CS, Larsen L, Wiese L, Dalager-Pedersen M, Claggett BL, Janstrup KH, Duran-Parrondo C, Pineiro-Sotelo M, Cribeiro-Gonzalez M, Conde-Pajaro M, Miras-Carballal S, Gonzalez-Perez JM, Solomon SD, Sivapalan P, Martel CJ, Jensen JUS, Martinon-Torres F, Biering-Sorensen T; DANFLU-2 Study Group; GALFLU Trial Team. Effectiveness of high-dose influenza vaccine against hospitalisations in older adults (FLUNITY-HD): an individual-level pooled analysis. Lancet. 2025 Nov 22;406(10518):2425-2434. doi: 10.1016/S0140-6736(25)01742-8. Epub 2025 Oct 17. PMID 41115437